CLINICAL TRIAL: NCT06768190
Title: WhatsApp-based Psycho-socio-educational Intervention (WeLove) for Prevention of Psychological and Sleep Problems in Pregnant Women and Their Partners: A Three-arm Double-blinded Pilot Randomised Controlled Trial
Acronym: WhatsApp-based
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Hospital Authority, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Lau Ying, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RS-2023-LY
Record Dates: First submitted 2024-12-31; First posted 2025-01-10 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Sleep Problems; Psychological; Well-Being, Psychological
Keywords: Couple-based intervention; Psycho-socio-educational intervention (WeLove); Psychological well-being; Sleep outcome
MeSH Terms: conditions — Parasomnias; Psychological Well-Being | interventions — Family Characteristics

STUDY DESIGN:
Intervention Model Description: Double-blinded Pilot
Who Masked: Participant, Outcomes Assessor
Masking Description: The randomization of participants will enable the enrolling researcher to remain blind to participant conditions throughout the trial. The research assistants evaluating the participants are blinded to the group assignment. The assistants analysing participant data are also blinded to the group assignment. The active nature of the control condition may also allow us to blind the participants to the condition. The participants will be informed that the study aims to investigate the efficacy of three conditions to improve psychological and sleep well-being. However, they will not be explicitly advised of the content or intention. This minor deception is designed to yield a double-blind trial of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention group 1 (Experimental): In intervention group 1, pregnant women and their partners will participate in a six-week Welove intervention. The intervention comprises six sessions, including psychoeducation, communication training, sleep hygiene, stimulus control, cognitive restructuring, and behavioural activation.
  Interventions: Behavioral: WhatsApp-based psycho-socio-educational intervention (WeLove)
- Intervention group 2 (Experimental): In intervention group 2, only pregnant women will participate in a six-week WeLove intervention. The intervention comprises six sessions, including psychoeducation, communication training, sleep hygiene, stimulus control, cognitive restructuring, and behavioural activation.
  Interventions: Behavioral: WhatsApp-based psycho-socio-educational intervention (WeLove)
- Control (Placebo Comparator): In the control group, pregnant women and their partners are instructed to use WhatsApp as normal for six weeks.
  Interventions: Behavioral: WhatsApp as usual

INTERVENTIONS:
Behavioral: WhatsApp as usual — Pregnant women and their partners are instructed to use WhatsApp as normal for six weeks.
  Other Names: WhatsApp for couple
  Arms: Control
Behavioral: WhatsApp-based psycho-socio-educational intervention (WeLove) — The intervention comprises six sessions, including psychoeducation, communication training, sleep hygiene, stimulus control, cognitive restructuring, and behavioural activation. Each session has two short videos, quizzes, forums, and homework. The content is presented through a virtual midwife using storytelling of real-life scenarios, animation, and case vignettes about psychological and sleep problems during pregnancy. A virtual midwife acts as an educator to explain the prevalence, causes, and factors of psychological and sleep problems. Every session will concentrate on certain courses and offer specialised advice to expectant mothers and their partners. Using the security links on the WhatsApp platform, each session takes 15 to 20 minutes to finish.
  Arms: Intervention group 1; Intervention group 2

SUMMARY:
Objectives: (1) evaluate the feasibility and acceptability of the WhatsApp-based psycho-socio-educational intervention (WeLove); (2) preliminarily examine the effects of the intervention on psychological symptoms (depression, anxiety, stress symptoms), sleep quality, and life satisfaction; and (3) preliminarily examine the interdependence between psychological symptoms and sleep quality in pregnant women and their partners.

Methods: The investigators will use WhatsApp to provide the six sessions of the intervention, which include psychological, social, and educational components. A three-arm double-blinded pilot randomised controlled trial (RCT) is used in 60 couples, followed by individual face-to-face interviews for process evaluation in 10 to 20 couples based on data saturation. Participants will be assigned to one of three groups and 20 couples per group: intervention 1 (couples for WeLove), intervention 2 (pregnant women for WeLove), or the control group (use WhatsApp as normal). Participants will be assessed pre- and post-intervention. Generalised estimating equation analysis and thematic analysis will be performed to examine the research objectives.

DETAILED DESCRIPTION:
Study design A prospective randomised double-blind, three-arm, parallel-group design will be adopted. The report of the trial will follow the Consolidated Standards of Reporting Trials guidelines for an Internet-based intervention (CONSORT-EHEALTH).

ELIGIBILITY:
Inclusion Criteria:

* pregnant with a gestation of >12 to 28 weeks and their partners over 18 years
* able to read and understand Chinese
* have electronic devices with WhatsApp that can contact the Internet
* can provide written consent and voluntary participation in this study

Exclusion Criteria:

* current severe medical illnesses
* psychological and sleep disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Psychological outcome: Depression, anxiety and stress symptoms | Baseline, pre-intervention and immediately after the intervention
  Depression, anxiety and stress symptoms will be assessed by the Chinese version of 21-item Depression Anxiety and Stress Scale (DASS-21). It has three subscales with seven items each: stress, anxiety, and depressive symptoms. Four-point rating scales, ranging from 0 (did not apply to me at all) to 3 (applied to me very much or most of the time), are used to categorise frequency and severity. The final scores are obtained by multiplying each subscale's values by two. Every subscale has a total score that varies from 0 to 42; a high score on any subscale denotes a higher level of stress, anxiety, and depressive symptoms

SECONDARY OUTCOMES:
Sleep outcomes: Subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, sleep medication, and daytime dysfunction | Baseline, pre-intervention and immediately after the intervention
  Subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, sleep medication, and daytime dysfunction will be assessed by the Chinese version of 19-item Pittsburgh Sleep Quality Index (PSQI). Subjective sleep quality, sleep latency, duration, habitual sleep efficiency, sleep disruptions, sleep medication, and daytime dysfunction are the seven components that comprise the components of the PSQI. The range of scores for each item is 0 (no difficulty) to 3 (extreme difficulty). The total score ranges between 0 and 21. Poorer quality of sleep is indicated by a higher overall score
Psychological well-being: Subjective well-being | Baseline, pre-intervention and immediately after the intervention
  Subjective well-being will be measured by the Chinese version of World Health Organization-Five Well-Being Index (WHO-5). It included 5 items. Each item is rated on a six-point Likert scale, ranging from 0 (at no time) to 5 (always), the total score range from 0 to 25. A higher score indicates greater mental well-being.

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
The data collection is not start yet and our research team does not decide the plan to share data.